CLINICAL TRIAL: NCT06628570
Title: Screening Strategies Among High-risk Populations for Anal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lisa Flowers (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Lisa Flowers, Professor of Medicine, Emory University
Organization: Emory University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY00006091; R01CA285198 (NIH)
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms; HPV-Related Anal Squamous Cell Carcinoma
Keywords: Cancer; HIV; Screening
MeSH Terms: conditions — Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Men with impaired immune status (Other): At each study visit, participants will receive a digital anorectal examination followed by HRA, with directed biopsies of suspicious lesions. An HRA-certified physician will collect anal swabs and HRA-directed biopsies for histological confirmation of disease and biomarker assays.
  Interventions: Diagnostic Test: HRA + Biopsy; Diagnostic Test: Anal Cytology; Diagnostic Test: Genotyping of anal hrHPV infection; Diagnostic Test: CINtec®PLUS
- Men without impaired immune status (Other): At each study visit, participants will receive a digital anorectal examination followed by HRA, with directed biopsies of suspicious lesions. An HRA-certified physician will collect anal swabs and HRA-directed biopsies for histological confirmation of disease and biomarker assays.
  Interventions: Diagnostic Test: HRA + Biopsy; Diagnostic Test: Anal Cytology; Diagnostic Test: Genotyping of anal hrHPV infection; Diagnostic Test: CINtec®PLUS
- Women with impaired immune status and high grade LGTN (Other): At each study visit, participants will receive a digital anorectal examination followed by HRA, with directed biopsies of suspicious lesions. An HRA-certified physician will collect anal swabs and HRA-directed biopsies for histological confirmation of disease and biomarker assays.
  Interventions: Diagnostic Test: HRA + Biopsy; Diagnostic Test: Anal Cytology; Diagnostic Test: Genotyping of anal hrHPV infection; Diagnostic Test: CINtec®PLUS
- Women without impaired immune status with high grade LGTN (Other): At each study visit, participants will receive a digital anorectal examination followed by HRA, with directed biopsies of suspicious lesions. An HRA-certified physician will collect anal swabs and HRA-directed biopsies for histological confirmation of disease and biomarker assays.
  Interventions: Diagnostic Test: HRA + Biopsy; Diagnostic Test: Anal Cytology; Diagnostic Test: Genotyping of anal hrHPV infection; Diagnostic Test: CINtec®PLUS

INTERVENTIONS:
Diagnostic Test: HRA + Biopsy — High-Resolution Anoscopy, or HRA, is a standard of care procedure for screening and detection of premalignant lesions of the anus. Using a small, thin round tube called an anoscope, the anal canal is examined with a high-resolution magnifying instrument called a colposcope. The application of a mildly acidic liquid on the anal canal facilitates the evaluation of abnormal tissue such as anal dysplasia. Biopsies for histological confirmation of disease will be taken. Biopsies' reporting will follow the terminology, criteria, and recommendations of the Lower Anogenital Squamous Terminology (LAST) project. Histology results will be reported as benign, condyloma acuminatum, AIN grades 1-3, or cancer. For the proposed project, aHSIL+ will be defined as AIN2 (p16 block-positive), AIN3, and cancer at the HRA encounter. All other cases will be classified as <aHSIL, including benign, condyloma acuminatum, and AIN1
  Other Names: HRA and Histology
Diagnostic Test: Anal Cytology — Anal cytology collection (swab samples) will be performed as part of the standard of care during this study. The collected cells, suspended in the SurePath liquid-based medium, will be placed on a slide and microscopically examined by a board-certified pathologist. The sample will then be interpreted using the Bethesda System: negative for intraepithelial lesion or malignancy (NILM), ASCUS, LSIL, ASC-H, or HSIL. Pathologists interpreting the anal cytology will be blinded from hrHPV testing and biopsy histology.
  Other Names: Swab anal Sample
Diagnostic Test: Genotyping of anal hrHPV infection — Samples of exfoliated cells from the anal canal will be collected with Dacron swabs. To identify the infecting HPV genotype, DNA will be extracted from swab samples collected with the MagNA Pure LC DNA Isolation Kit III and an LC MagNA Pure system (Roche Diagnostics GmbH, Mannheim, Germany), followed by HPV typing using the TypeSeq assay, a laboratory prepared high-throughput next-generation sequencing assay developed by NCI will be performed as described. The assay uses three sequential PCR steps resulting in barcoded L1 amplicons sequenced and submitted to a bioinformatics pipeline for typing. This TypeSeq assay qualitatively detects and identifies 51 HPV genotypes (HPV types 3, 6, 11, 13, 16, 18, 26, 28, 30, 31, 32, 33, 34, 35, 39, 40, 42, 43, 44, 45, 51, 52, 53, 54, 56, 58, 59, 61, 62, 66, 67, 68, 69, 70, 71, 72, 73, 74, 76, 81, 82, 83, 84, 85, 86, 87, 89, 90, 91, 97, and 114), including 14 high-risk (16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 68)
  Other Names: hrHPV
Diagnostic Test: CINtec®PLUS — Samples of exfoliated cells from the anal canal will be collected with Dacron swabs. Dual immunostaining with p16/Ki-67 will be performed on the residual cytologic specimen by Roche MTM Laboratories (Heidelberg, Germany), using the CINtec®PLUS Kit according to the manufacturer's instructions. The anal cytology material will be stained with a mouse monoclonal antibody directed against human p16INKa (p16) protein (clone E6H4) and recombinant rabbit monoclonal antibody directed against human Ki-67 protein (clone 274-11AC3V1), using the BenchMark ULTRA instrument (Ventana Roche). Samples with insufficient cellularity will be excluded from the evaluation. A trained cytotechnologist will review all cases for cells staining positively with both markers. A slide will be considered positive if 1 or more squamous epithelial cell(s) stained positive for both p16 and Ki-67 and dual stain-positive cells will be semi-quantitatively assessed (0, 1, 2-5, 6-50, >50).
  Other Names: P16/Ki-67 dual immunostaining

SUMMARY:
The goal of the proposed research is to 1) examine the performance of emerging screening methods for anal high-grade squamous intraepithelial lesion (aHSIL), a precancerous condition of anal cancer, among populations at high risk for anal cancer and 2) characterize DNA methylation, immunologic response, and environmental factors associated with aHSIL.

DETAILED DESCRIPTION:
Anal cancer, caused by persistent infection with high-risk human papillomavirus (hrHPV), is typically preceded by anal high-grade squamous intraepithelial lesions (aHSIL). The incidence and mortality of advanced anal cancer has been increasing in the U.S., with the greatest burden of disease and mortality in individuals with chronic impairment of the immune system. The study is important because the incidence of anal cancer is particularly high among certain groups. Findings will provide much-needed evidence for anal cancer screening strategies to reduce incidence of anal cancer and improve health outcomes. The study population includes individuals with chronic impairment of the immune system and females with a known history of high-grade lower genital tract neoplasia.

The study procedures include filling out self-reported questionnaires and collecting biosamples for study-related assays. HRA is part of the standard clinic procedure for this group of participants. Collected biosamples will be banked for future research use. In-person or remote signed consent may occur for the study.

ELIGIBILITY:
Inclusion Criteria:

* 30-80 years of age
* Individuals with chronic impaired immune status
* History of high-grade lower genital tract neoplasia (LGTN), Zubrod Performance Status of 0-2;

Exclusion Criteria:

* Patients treated for aHSIL less than 6 months before screening,
* History of anal cancer and pregnant women.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Specificity and Sensitivity of screening markers | Baseline
  Sensitivity and specificity will be calculated for each of the proposed screening markers separately and a combination of two and three markers for the detection of aHSIL at baseline. The combination of the two and three markers of primary interest includes CINtec®PLUS +hrHPV, CINtec®PLUS+anal cytology, hrHPV+anal cytology, and CINtec®PLUS+hrHPV+anal cytology. The analysis will be performed for the four high-risk groups together and stratified by the four high-risk categories.

SECONDARY OUTCOMES:
DNA methylation markers | Baseline, 1 year, 2 years
  In these models, aHSIL status at baseline will be considered as the response, and each anal DNA methylation marker will be the predictor. Separate models will be performed for each methylation marker (ZNF582, ASCL1, ZIC1, SST, LHX8, WDR17, and ST6GALNAC5)
Anal immune modulations | Baseline, 1 year, 2 years
  High-risk HPV 16 persistent patients (N=10) vs. patients with no HPV at least two consecutive times (N=10). Each of the groups will also include aHSIL+ (N=5) vs. <aLSIL (N=5).
aHSIL prevalence | Baseline
  The prevalence of HSIL will be estimated as the proportion of participants who are HRA positive for HSIL at entry and its 95% confidence interval. Logistic regression analysis will be used to evaluate the association of potential risk factors with diagnosis of HSIL.
aHSIL clearance | 1 year, 2 years
  Only people treated with aHSIL will be used for the clearance analysis. Clearance (HRA biopsy-proven) will be defined as no detectable aHSIL at the immediate one-year (for those with baseline aHSIL) or two-year (for those with newly diagnosed aHSIL cases at the one-year visit) follow-up visit after aHSIL treatment.
Inflammatory Markers (Il-1RA, IL1β, IL6, IL6sr, TNF-α, and IL-10) | Baseline, 1 year, 2 years
  Anal swab concentrations of inflammatory markers (IL1ra, IL1β, IL6, IL6sr, TNF-α, and IL-10) will be determined using multiplex assays (Meso Scale Discovery, Rockville, MD) according to the manufacturer's protocol. All samples will be run in duplicates, and mean intra- and inter-assay CVs will be calculated and expected to be <10%. These inflammatory markers have been reliably found to be elevated in inflammatory-associated diseases including anal inflammation.
Inflammatory Markers (sTNFR2 and interferon (IFN)-γ) | Baseline, 1 year, 2 years
  Anal swab concentrations of inflammatory markers of inflammatory markers (sTNFR2 and interferon (IFN)-γ) will be determined using multiplex assays (Meso Scale Discovery, Rockville, MD) according to the manufacturer's protocol.
Inflammatory Marker (CRP) | Baseline, 1 year, 2 years
  Anal swab concentrations of inflammatory markers (CRP) will be determined using multiplex assays (Meso Scale Discovery, Rockville, MD) according to the manufacturer's protocol. All samples will be run in duplicates, and mean intra- and inter-assay CVs will be calculated and expected to be <10%.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flowers, MD, MPH, Principal Investigator — Emory University; Canhua Xiao, PhD, RN, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - University of Miami School of Medicine at Jackson Memorial Hospital (JMH), Miami, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - The Ponce Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected from study participation will be available for sharing after deidentification
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available for sharing after publication.
Access Criteria: Data will be shared upon request with researchers who provide a methodologically sound proposal to achieve the aims in the approved proposal. To gain access, data requesters will need to sign a data access agreement.